CLINICAL TRIAL: NCT04665102
Title: Validation of a Transfer Learning Deep Learning Algorithm for Image Classification in Multiple Pathologies
Brief Title: Pilot Study on Deep Learning in the Eye
Acronym: IDLE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CRG UZ Brussel (Other)
Responsible Party: Principal Investigator, Pieter Nelis, Researcher, CRG UZ Brussel
Other Study IDs: IDLE1000
Record Dates: First submitted 2020-12-07; First posted 2020-12-11 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Central Serous Chorioretinopathy; Diabetic Retinopathy; Cataract
MeSH Terms: conditions — Central Serous Chorioretinopathy; Diabetic Retinopathy; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- No pathology
- Pathology
  Interventions: Other: Image classification using deep learning algorithm

INTERVENTIONS:
Other: Image classification using deep learning algorithm — Image classification using deep learning algorithm
  Groups: Pathology

SUMMARY:
Deep learning allows you to classify images using a self-learning algorithm. Transfer learning builds on an existing self-learning algorithm to enable image classification with fewer images. In this study, this technique will be applied to different image modalities in different syndromes. Retrospective study design.

ELIGIBILITY:
Inclusion Criteria:

* Availability of images, which allow discrimination.

Exclusion Criteria:

* No availability of clear data on disease differentiation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy and non-healthy subjects: extract data out of available images
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Validation of Image classification by transfer learning algorithm | 1 year

IPD SHARING:
Plan to Share IPD: No